CLINICAL TRIAL: NCT06724185
Title: Effects of LP28 on Immunity Enhancement in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synbio Tech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SF24108C
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Common Cold; Immunity; Probiotic
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LP28 capsule (Experimental): Subjects will take two capsule of the experimental group(LP28 capsule) within 30 minutes before breakfast and dinner each day.
  Interventions: Dietary Supplement: LP28 capsule
- Placebo capsule (Placebo Comparator): Subjects will take two placebo capsule within 30 minutes before breakfast and dinner each day.
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: LP28 capsule — LP28 capsule : 5.0×10^9 CFU/capsule
  Arms: LP28 capsule
Dietary Supplement: Placebo Capsule — Maltodextrin
  Arms: Placebo capsule

SUMMARY:
Due to the increasing attention on aging-related health issues, this study focuses on the elderly population as participants. The aim is to investigate whether supplementation with Lactobacillus plantarum LP28 can effectively enhance immunity, reduce the frequency and severity of common cold infections, and ultimately promote overall health in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Those who had symptoms of common cold or tonsillitis at least twice in the past year.

Exclusion Criteria:

* People who have liver, kidney, immune, or neoplastic diseases diagnosed by doctor.
* People with mental illnesses such as schizophrenia or depression.
* People who have allergic rhinitis.
* People who have a current condition of drug or alcohol dependence.
* Any person is deemed inappropriate by the researcher for the clinical trial.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
WURSS-24 | From enrollment to the end of treatment at 12 weeks (measure daily)
  The WURSS-24 (Wisconsin Upper Respiratory Symptom Survey-24) is a questionnaire designed to assess the impact of upper respiratory tract infections, such as the common cold, on daily life and health. It includes 24 questions covering symptoms (e.g., cough, runny nose, fatigue) and how they affect daily activities, work, and social interactions. Patients rate each item on a scale from 0 (no problem) to 7 (severe problem).

SECONDARY OUTCOMES:
Immune cell ratio | From enrollment to the end of treatment at 12 weeks (measure every 6 weeks)
  Blood samples were collected, and the proportions of immune cells were analyzed using flow cytometry, including: (1) CD3+/lymphocyte, (2) CD4+/CD3+, (3) CD8+/CD3+, and (4) CD56+CD16+/lymphocyte.
NK cell activity | From enrollment to the end of treatment at 12 weeks (measure every 6 weeks)
  Peripheral blood mononuclear cells (PBMCs) were isolated, and magnetic bead-based separation was used to deplete non-NK cells. The K562 human immortalized myelogenous leukemia cell line was then used as target cells, and the proportion of K562 cells lysed by NK cells was measured as an indicator of NK cell activity.
Cytokines measurement | From enrollment to the end of treatment at 12 weeks (measure every 6 weeks)
  Plasma was collected, and cytokine concentrations were analyzed using enzyme-linked immunosorbent assay (ELISA). The detection items included IL-4, IL-6, IL-12, IFN-γ, CRP and TNF-α.
sIgA | From enrollment to the end of treatment at 12 weeks (measure every 6 weeks)
  Saliva samples were collected, and Secretory immunoglobulin A (sIgA) concentrations were analyzed using enzyme-linked immunosorbent assay (ELISA).
α-amylase | From enrollment to the end of treatment at 12 weeks (measure every 6 weeks)
  Saliva samples were collected, and α-amylase concentrations were analyzed using enzyme-linked immunosorbent assay (ELISA).
GSRS questionnaire | From enrollment to the end of treatment at 12 weeks (measure weekly)
  The Gastrointestinal Symptom Rating Scale (GSRS) is a questionnaire used to evaluate the severity of gastrointestinal symptoms. It includes questions on five key areas: abdominal pain, reflux, diarrhea, indigestion, and constipation. Patients rate their symptoms on a 7-point Likert scale, where higher scores indicate more severe symptoms.
Defecation frequency and stool pattern | From enrollment to the end of treatment at 12 weeks (measure weekly)
  Defecation frequency was recorded, and stool characteristics, including shape, consistency, and color, were documented using the Bristol Stool Chart.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Chung Hsing University, Taichung
  - Taichung Veterans General Hospital, Taichung